CLINICAL TRIAL: NCT06798155
Title: Effect of Listening to Standardized Music Sequences on Preventing Postoperative Pain in Proctologic Surgery
Acronym: MUSICOPROCTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint-Vincent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24.04190.000403
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Hemorrhoid; Anal Fistulas; MUSICAL THERAPY; Anal Fissure and Fistula
Keywords: Standardized Music Therapy; Proctologic Surgery; Pain Management; Analgesic Use; Randomized Controlled Trial; Music Intervention; Preoperative Care; Monocentric Study
MeSH Terms: conditions — Hemorrhoids; Rectal Fistula; Fissure in Ano; Fistula; Agnosia

STUDY DESIGN:
Intervention Model Description: The design of this study does not fall within the framework of a specific phase but rather corresponds to a Category 2 study under the Jardé law. In other words, it qualifies as a RIPH2 study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized Music Listening (Experimental): Participants assigned to this arm will benefit from standardized music listening sessions via the Music Care® application.
  Pre-surgery: At the entrance to the operating room, participants will spend 20 minutes lying on a stretcher in a dedicated room, listening to relaxing music sequences through a tablet and headphones provided by the research team. Participants can select their preferred musical style, tempo, and tracks.
  Post-surgery: Participants will continue listening to music sequences daily for 20 minutes at home using their own devices (smartphone, tablet, or computer) until day 28 post-surgery.
  Interventions: Other: Standardized Music Listening Therapy
- Standard Care (No Intervention): Participants assigned to this arm will not benefit from standardized music listening sessions.
  Pre-surgery: Participants will proceed directly from their hospital room to the operating room without a music listening session.
  Post-surgery: Participants will be managed according to standard care practices, with no additional interventions related to music therapy.

INTERVENTIONS:
Other: Standardized Music Listening Therapy — Type of Intervention: Pre- and postoperative listening to standardized music sequences designed specifically for relaxation and pain management.
  Delivery Method: Sessions are conducted via the Music Care® application, using a tablet and headphones provided during hospitalization. Participants select their preferred music style, tempo, and tracks to tailor the experience to their preferences.
  Duration and Schedule:
  Pre-surgery: One 20-minute session in a dedicated room before entering the operating theater.
  Post-surgery: Daily 20-minute sessions at home for 28 days post-surgery using participants' own devices (smartphone, tablet, or computer).
  Purpose: To evaluate the effect of music on reducing postoperative pain, minimizing analgesic use, and improving the quality of life.
  Distinctiveness: This intervention uniquely integrates patient-controlled music preferences with a structured listening regimen before and after surgery, offering a personalized approach to enhancing recovery outcom
  Arms: Standardized Music Listening

SUMMARY:
The study, "Effect of Listening to Standardized Music Sequences on Preventing Postoperative Pain in Proctologic Surgery," aims to evaluate the impact of preoperative listening to standardized music sequences on postoperative pain in patients undergoing proctologic surgery (for hemorrhoids, fistulas, or anal fissures).

This research will assess the influence of preoperative music on postoperative pain management, the use of analgesics after surgery and during the following month, and its effect on the quality of life post-surgery.

MUSICO-PROCTO is an interventional, randomized study involving two groups (patients will be randomly assigned to either the music intervention or control group). The study is monocentric, conducted at Clinique Saint Vincent in France, and includes 550 participants.

Participants will be followed for 28 days, while the overall study duration will span 28 months.

To participate, individuals must:

Be aged 18 or older. Be affiliated with a social security system. Provide signed informed consent. Undergo proctologic surgery for hemorrhoids, fistulas, or anal fissures. This study seeks to explore the potential of music as a complementary method to improve postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged over 18 years.
* Patient who has signed an informed consent form.
* Patient scheduled to undergo proctological surgery (for hemorrhoids, fistula, or anal fissure) at the participating institution.
* Must be affiliated with a social security system or be a beneficiary of such a system.
* Patient must have access to the necessary technical means (smartphone, computer, tablet) to use the Music Care® application.

Exclusion Criteria:

* Refusal to consent.
* Patient unable to read, write, or understand French.
* Vulnerable patient according to Article L1121-6 of the French Public Health Code (CSP).
* Adult patient under guardianship or curatorship or under legal protection (safeguard of justice).
* Patient unable to personally give informed consent according to Article L.1121-8 of the CSP or an adult protected by law.
* Pregnant or breastfeeding women according to Article L1121-5 of the CSP.
* Patient who has already participated in a study within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (EVA Pain) in the recovery room (SSPI). | Immediately post-surgery in the recovery room.
  First postoperative pain measurement using the EVA (Visual Analog Scale), scored from 0 to 10, in the recovery room (SSPI).

SECONDARY OUTCOMES:
Successive Pain and Anxiety Scores (EVA Pain and EVA Anxiety) | From hospitalization to Day 28 post-surgery.
  Successive measurements of pain and anxiety using the EVA scales, scored from 0 to 10, at the following time points:
  Admission to hospitalization. 30 minutes after premedication. In the recovery room (SSPI). At hospital discharge. Day 10 (±3 days). Day 28 (follow-up visit).
State Anxiety Score (STAI-Y-ETAT) | From hospitalization to Day 28 post-surgery.
  Evaluation of state anxiety using the STAI-Y-ETAT scale at the following time points:
  Admission to hospitalization. 30 minutes after premedication. At hospital discharge. Day 28 (follow-up visit)
Kess Score | From hospitalization to Day 28 post-surgery
  Measurement of bowel function using the Kess score at the following time points:
  Admission to hospitalization. 30 minutes after premedication. Day 10 (±3 days). Day 28 (follow-up visit).
Total Time in SSPI and Hospitalization Duration | During the hospital stay.
  Measurement of the total time spent in the recovery room (SSPI) and overall hospitalization duration.
Total Analgesic Consumption During Hospital Stay | Measured from hospital admission to hospital discharge, within an estimated time frame of 6 to 24 hours (due to the outpatient nature of the procedure).
  The total amount of analgesic medication consumed during the entire hospital stay.
Time to Healing | From surgery to Day 28 post-surgery.
  Measurement of wound healing time by assessing wound surface area using the Imito Measure application, in the genu-pectoral position.
Quality of Life Scores (HEMO-FISS-QoL and EQ5D-5L) | From hospitalization to Day 28 post-surgery.
  Assessment of quality of life using the HEMO-FISS-QoL and EQ5D-5L scales at the following time points:Admission to hospitalization.
  Day 28 (follow-up visit).
Patient Satisfaction | Immediately post-surgery, upon discharge from SSPI.
  Measurement of patient satisfaction using a Likert scale upon discharge from the recovery room (SSPI).
Medico-Economic Impact | During the hospital stay.
  Assessment of the economic impact of the intervention by recording:
  Operative times. Recovery room durations. Total hospitalization duration (in minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint Vincent, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.music.care/